CLINICAL TRIAL: NCT07043920
Title: The Association Between Daily Physical Activity Level and Nicotine Dependence in University Students: A Cross-Sectional Study
Brief Title: Impact of Smoking on Physical Activity Level in Young Adults
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: FA-Nosmoke-1
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Smoking Behaviors; Physical Inactivity
MeSH Terms: conditions — Smoking; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoker Group: This group will consist of university students aged 18 years and older who report currently smoking cigarettes on a regular basis. Their level of nicotine dependence will be assessed using the Fagerström Test for Nicotine Dependence (FTND). They will also complete the International Physical Activity Questionnaire-Short Form (IPAQ-SF) to evaluate their weekly physical activity levels.
  Interventions: Other: Behavioral Assessment (No therapeutic intervention will be administered)
- Non-Smoker Group: This group will include university students aged 18 years and older who have never smoked or used tobacco products. Their physical activity levels will be assessed using the IPAQ-SF. FTND will not be applied as they have no smoking history.
  Interventions: Other: Behavioral Assessment (No therapeutic intervention will be administered)

INTERVENTIONS:
Other: Behavioral Assessment (No therapeutic intervention will be administered) — Participants will complete two validated questionnaires:
  The Fagerström Test for Nicotine Dependence (FTND) - to assess levels of nicotine dependence.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) - to quantify weekly physical activity levels (walking, moderate, vigorous).

SUMMARY:
This study will aim to examine the relationship between the daily physical activity level and nicotine dependence severity in university students. By identifying whether a higher physical activity level is associated with lower levels of smoking, the findings will help inform interventions to support healthier lifestyles in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Studying in a health-related university program
* Healthy individuals (no known chronic disease)
* Voluntarily agreeing to participate

Exclusion Criteria:

* History of cardiovascular disease, cancer, or severe respiratory illness
* Pregnancy
* Age under 18

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Participants will consist of healthy university students aged 18 years and older, studying in health sciences departments in Istanbul, Türkiye. Both smokers and non-smokers will be included. Participants with cardiovascular disease, cancer, chronic pulmonary conditions, or pregnancy will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Total physical activity score | At baseline (single timepoint)
  Total weekly physical activity will be assessed using International Physical Activity Score- Short Form (IPAQ-SF) and expressed as MET-min/week. Categories will be created as inactive, minimally active, and very active.

SECONDARY OUTCOMES:
Fagerström Test for Nicotine Dependence (FTND) | At baseline (single timepoint)
  The Fagerström Test for Nicotine Dependence (FTND) is a widely used, standardized, 6-item questionnaire designed to assess the intensity of physical addiction to nicotine. The test evaluates behaviors and patterns related to cigarette smoking, including time to first cigarette after waking, number of cigarettes smoked per day, and difficulty refraining from smoking in forbidden areas. Each item is scored, and the total score ranges from 0 to 10.
  Score 0-3: Low dependence
  Score 4-6: Moderate dependence
  Score 7-10: High dependence
  The FTND allows researchers and clinicians to categorize smokers according to their nicotine addiction level, which can be useful for tailoring interventions or for observational analysis of behavior and health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Turkey (Türkiye)